CLINICAL TRIAL: NCT05946655
Title: Evaluation of the Congruity of Methods Used in the Diagnostics of Chronic Endometritis in the Course of Infertility and the Effectiveness of Antibiotic Therapy in the Context of Remission of Symptoms and Obstetric Results
Brief Title: Diagnostics of Chronic Endometritis in Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, M.D., Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1072.6120.322.2020
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Infertility Unexplained; Abnormal Uterine Bleeding; Intrauterine Disorder
Keywords: Infertility Unexplained; Chronic endometritis; Office hysteroscopy; Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Ofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic therapy (Experimental): Women diagnosed with CE undergoing empirical antibiotic therapy
  Interventions: Drug: Ofloxacin + Metronidazole
- Control (No Intervention): Women diagnosed with CE not subjected to empirical antibiotic therapy

INTERVENTIONS:
Drug: Ofloxacin + Metronidazole — Ofloxacin 2x200mg orally for 10 days + Metronidazole 1x500 mg vaginally for 10 days
  Arms: Antibiotic therapy

SUMMARY:
Chronic endometritis (CE) is characterized by the presence of atypical plasma cell infiltrates (CD138 positive) in the endometrial stroma. Recent analyzes suggest that CE adversely affects fertility by reducing endometrial receptivity, impairing decidualization and uterine contractility, thus increasing the risk of recurrent pregnancy loss and implantation failure. It is likely that a significant proportion of idiopathic infertility cases are due to CE. The diagnosis of CE is a challenge because the clinical examination and transvaginal ultrasonography are considered non-specific. The recent scientific research has been aimed at identifying hysteroscopic CE diagnostic criteria and establishing the compatibility of ultrasonographic, hysteroscopic, histopathological (including the use of immunohistochemical testing with antibodies against human CD138) and microbiological diagnoses. Preliminary literature results suggested that successful treatment of CE with antibiotics could improve live birth rates.

DETAILED DESCRIPTION:
The objectives are as follows:

1. Estimation of the diagnostic congruity of hysteroscopic, histopathological and microbiological diagnoses of CE
2. Estimation of the effectiveness of empirical antibiotic therapy in the treatment of CE, confirmed by normalization of the hysteroscopic appearance of the uterine cavity, normalization of histopathological results of endometrial biopsies and decrease in plasma cell count/1 high power field (HPF)
3. Estimation of the percentage of clinical pregnancies achieved in women subjected to empiric antibiotic therapy for CE vs. in women without treatment. The study group will consist of women of childbearing age subjected to office hysteroscopy due to intrauterine pathologies, AUB, and idiopathic infertility. The prerequisite for hysteroscopy is a normal cervical cytology result, a negative blood pregnancy test, a normal vaginal biocenosis and the first phase of the cycle. During hysteroscopy, the following will be performed: visual inspection of the uterine cavity in search of focal lesions and features of the endometrium suggestive of CE, such as: focal or diffuse hyperemia, micropolyps, stromal edema, then collection of washings from the uterine cavity for microbiological examination (aerobic and anaerobic culture, PCR for Chlamydia, culture for Mycoplasma, Ureaplsma) and excision of the focal lesion or endometrial biopsy. The extracted tissue material will be subjected to standard histopathological examination with hematoxylin and eosin staining. Additional immunohistochemical staining with Monoclonal Mouse Anti-Human CD138 antibodies will be used to detect plasmocytes. The cut-off point for the number of CE-defining plasmocytes will be determined by the Receiver Operating Characteristic (ROC) curve. Women diagnosed with CE will be assigned to 2 arms: 1) ofloxacin 2x200 mg orally for 10 days + metronidazole 1x500 mg vaginally for 10 days, 2) control arm (no treatment). In the third cycle after the primary hysteroscopy, women will undergo a follow-up office hysteroscopy for a visual assessment of the uterine cavity and a follow-up endometrial biopsy. The percentage of women with improvement in the clinical appearance of the uterine cavity, normalization of histopathology and persistent CE in both arms will be determined. Data will be obtained on the results of infertility treatment (obtaining a clinical pregnancy) within 24 months of the procedure or completion of antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* lack of previous diagnosis and treatment due to suspected pathology of the uterine cavity
* lack of active infection of the reproductive tract

Exclusion Criteria:

* pelvic surgery performed within 6 months preceding the hysteroscopy
* confirmed pelvic endometriosis
* antibiotic or probiotic treatment within 3 months preceding the hysteroscopy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Determination of the cut-off point of the number of plasma cells/1 HPF corresponding to histological CE | 3 months
  Diagnostic compatibility assessment of immunohistochemistry and histopathology will be performed to estimate the cut-off point for the number of plasma cells defining CE using the ROC (Receiver Operating Characteristic) curve

SECONDARY OUTCOMES:
Assessment of the reliability of polyp visualization in diagnosing CE | 3 months
  The percentage of women with CE and a hysteroscopy-visible endometrial polyp and without a polyp will be calculated and compared
Assessment of the reliability of the visualization of focal endometrial hyperemia in the diagnosis of CE | 3 months
  The percentage of women with CE and hysteroscopy-visible focal hyperemia and without hyperaemia will be calculated and compared
Assesment of the reliability of the visualization of diffuse endometrial hyperemia in the diagnosis of CE | 3 months
  The percentage of women with CE and hysteroscopy-visible diffuse hyperaemia and without hyperaemia will be calculated and compared
Assessment of the reliability of the visualization of endometrial micropolyps in the diagnosis of CE | 3 months
  The percentage of women with CE and hysteroscopy-visible micropolyps and without micropolyps will be calculated and compared
Assessment of the reliability of the visualization of endometrial edema in the diagnosis of CE | 3 months
  The proportion of women with CE and hysteroscopy-visible endometrial edema and without endometrial edema will be calculated and compared
Evaluation of the effectiveness of antibiotic therapy in the context of reducing the number of plasma cells/1 mm2 | 3 months
  The number of plasma cells/1 mm2 will be calculated and compared among women who received antibiotic therapy in the course of CE and untreated women
Evaluation of the effectiveness of antibiotic therapy in the context of visual normalization of the uterine cavity in follow-up hysteroscopy | 3 months
  The percentage of women with persistent hysteroscopic CE symptoms: visualization of focal hyperemia or diffuse hyperemia or endometrial micropolyps or endometrial edema in follow-up hysteroscopy will be assessed and compared among women who received antibiotic therapy in the course of CE and untreated women
Evaluation of the effectiveness of antibiotic therapy in the context of normalization of histopathological results of a control endometrial biopsy | 3 months
  The percentage of women with persistent histopathological CE symptoms: presence of plasma cells and/or other inflammatory cells (lymphocytes or neutrophilic granulocytes or histiocytes/macrophages or eosinophilic granulocytes) destructing the endometrial tubuli among women who received antibiotic therapy in the course of CE and untreated women will be evaluated and compared in follow-up hysteroscopic endometrial biopsy
Evaluation of the effectiveness of antibiotic therapy in the treatment of CE - dependent infertility | 24 months
  Pregnancy rates will be assessed and compared among women who received antibiotics for CE and untreated women
Evaluation of the effectiveness of antibiotic therapy in the treatment of CE - dependent abnormal uterine bleeding | 24 months
  The rates of persistence of abnormal uterine bleeding will be assessed and compared in women who received antibiotics for CE and in untreated women.

OTHER OUTCOMES:
Evaluation of the frequency of isolation of a specific pathogen in the course of CE | 3 months
  The co-occurrence of a specific pathogen in CE and its type will be assessed using conventional microbiological methods

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., PhD, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No